CLINICAL TRIAL: NCT00169078
Title: A Study of the Impact of Insecticide-treated Curtains on the Prevalence of Antimalarial Drug Resistance in Children With Uncomplicated Malaria in Burkina Faso
Brief Title: Impact of Insecticide-treated Curtains on Antimalarial Drug Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITCR5093
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Transmission intensity; Insecticide-treated materials; antimalarial drug resistance
MeSH Terms: conditions — Malaria | interventions — Chloroquine

INTERVENTIONS:
Drug: Chloroquine

SUMMARY:
Attempts to understand the relationship malaria transmission intensity and antimalarial drug resistance had rested mainly on mathematical models. To date, except for two studies which reported reductions in the prevalence of drug resistance in Tanzania and Zimbabwe, no other field data addressed the impact of reducing malaria transmission by the use of vector control measures on antimalarial drug resistance. Thus whether vector control decrease or increase drug resistance remains a contentious issue. The aim of this study was to investigate the impact of insecticide-treated curtains (ITCs) on clinical and parasitological outcomes in children with uncomplicated malaria treated with chloroquine (CQ), on the prevalence of genetic markers of resistance to CQ and sulphadoxine-pyrimethamine (SP) and on the ability of children to clear drug resistant parasites. The therapeutic efficacy of CQ was studied in 9 villages which used ITCs for 6-8 years and 9 villages with no history of ITC use. A cross-sectional survey was also conducted to estimate the prevalence of genetic markers of resistance to CQ and SP in asymptomatic children.

DETAILED DESCRIPTION:
1. Background

   Drug resistance has been associated with increased numbers of hospital admissions, increased cases of clinical malaria and malaria-specific mortality . Several strategies have been proposed as means by which the spread of antimalarial drugs resistance could be delayed. These strategies include reducing drug pressure, improving the quality of drug use, using combinations of antimalarial drugs and use of vector control measures. Restricting the use of drugs to reduce drug pressure is presently unrealistic due to poor access to health facilities and a lack of equipment. Improving the quality of use of antimalarials through the use of pre-packaged doses, education and training is a sound control strategy. However, the impact of this strategy on drug resistance has not yet been evaluated. Another promising approach to contain drug resistance is the use of combination therapies. The most successful combinations so far are those using artemisinin and its derivatives. It is likely that implementing combination therapy in resource limited countries will be hampered by its high cost. Given their impact in reducing malaria transmission, cases of clinical malaria and all-cause malaria mortality, insecticide-treated materials (ITMs) have recently been proposed as a potential tool for delaying the development and spread of drug resistance. So far, the debate on the interaction between malaria transmission intensity and drug resistance has been driven by analytical models and, to our knowledge, only 2 field studies have yet addressed the impact of ITMs on antimalarial drug resistance. If ITMs reduced the development and spread of antimalarial drug resistance, this would enhance their usefulness as a malaria control tool. This study examines the impact of insecticide-treated curtains (ITC)used over 6-8 years on the prevalence of antimalarial drug resistance in Burkina Faso.
2. Objectives

   2.1 Primary objectives
   * To determine the frequency of in vivo clinical and parasitological failures following treatment of uncomplicated malaria with CQ in children living in villages protected and not protected by insecticide treated curtains (ITC).
   * To determine if children in ITC and non-ITC villages with clinical malaria differ in their ability to clear genetically resistant parasites after treatment with CQ.

   2.2 Secondary objectives
   * To determine the proportions of children infected with parasites carrying the pfcrt-76T and pfmdr1-86Y alleles associated with resistance to CQ in villages protected and not protected by ITC.
   * To determine the proportions of children infected with parasites carrying parasites with the dihydrofolate reductase (dhfr) and dihydropteroate synthetase (dhps) alleles associated with resistant to SP in ITC and non- ITC protected villages.
   * To relate in vivo clinical and parasitological failure rates to the presence of genotypic markers of resistance to CQ by estimating genotype-failure indices (GFIs) and genotype-resistance indices (GRIs).
3. Methods

3.1 Field work

Passive case detection was used to recruit children aged 6-59 months with uncomplicated malaria using a slightly modified version of the standard WHO in vivo method for assessing therapeutic efficacy of anti-malarial drugs .Children seeking care at the selected health centres were screened for eligibility to join the study, enrolled and followed up for 14 days. If a child's axillary temperature was >=37.5 ºC and no obvious cause of fever other than malaria was found on clinical examination, about 500 ml of blood was drawn into a micro-container containing EDTA. Microscopic diagnosis of malaria and measurement of packed-cell volume (PCV) were performed immediately after samples were received in the laboratory. After enrolment, further clinical examinations were performed on days 1, 2, 3, 7, and 14. In addition, the caretakers were advised to bring children back to the health centre at any time between day 1 and day 14 if the child's condition did not improve. Thick and thin blood films and filter paper blood spots were prepared on days 0, 3, 7, 14 and at unscheduled visits.

Treatment of children and treatment outcome

A standard treatment with CQ was administered to children with uncomplicated malaria. The treatment dosing was 25 mg/kg body weight of CQ over 3 days; 10 mg/kg on days 0, 1 and 5 mg/kg on day 2. Treatment was administered at the clinic under the supervision of a nurse. Outcomes for the in vivo trial were classified according to the WHO clinical and parasitological assessment system

Prevalence of pfcrt-76 and pfmdr1-86 mutations in the community

A cross-sectional survey was conducted to estimate the prevalence of pfcrt-76 and pfmdr1-86 mutations in asymptomatic children. Random samples of children aged 6 to 59 months and children aged 5 years to 14 years were selected per village. Thick and thin blood films and filter paper blood spots were prepared from a finger-prick.

Estimation of the entomological inoculation rate

A cross-sectional survey was conducted at the peak period of malaria transmission (September 2002) for the estimation of the EIR. Catches were performed using CDC light traps. An ELISA test was used to detect the presence of P. falciparum circumsporozoite protein (CSP).

Socio-economic and health seeking behaviour survey

In 2003, a survey was performed in a random sample of 20 compounds in each village to collect data on health seeking behaviour, socio-economic and demographic features of the study population including the frequencies of population movements between villages.

3.2 Laboratory methods

Thick and thin blood films were stained with Giemsa stain (3%) for 45 minutes. Asexual parasites and gametocytes of P. falciparum were counted against 400 white blood cells. For molecular biology analyses, DNA was extracted from pre, post-treatment and cross-sectional survey filter paper blood spots using chelex. DNA was amplified by nested PCR to detect mutations at pfcrt-76. Nest 2 PCR products were digested by Apo I endonuclease restriction enzyme and electrophoresed onto a 3% agarose. Sequence-specific oligonucleotide probing (SSOP) was performed to detect the presence of pfmdr1-86 mutation. Mutations at dhfr (51, 59 and 108) and at dhps ( 437 and 540) were also detected by SSOP. MSP2 gene polymorphisms were studied by PCR to differentiate recrudescence from new infections.

3.3 Sample size and power

With 18 communities (9 per group), the study would have 80% power to detect, at the 5% significance level, a 50% decrease in clinical failure rate in eligible children. This number of communities would also permit the detection of a 40% decrease in parasitological failure rate in eligible children with the same power, and at least 60% and 40% increases in clinical and parasitological failure rates, at 5% significance level, in children carrying parasites with CQ resistant genotypes before CQ treatment was started.

3.4 Data processing and analyses

Two data clerks independently entered data onto computers using EPIINFO version 6.0. Analyses were performed using STATA (Release 8.2, www.stata.com). The study main endpoints were examined using Generalized Estimating Equations regression model

3.5 Community approval

This was obtained after meetings with community leaders to explain the objectives of the study and what it involved. In addition to community consent, individual signed informed consent was obtained from caretakers of children before enrolment.

ELIGIBILITY:
Inclusion Criteria:

Age between 6 and 59 months Mono infection with P.falciparum malaria, with parasitaemia in the range of 1,000 to 150,000 parasites per ml Absence of danger signs or signs of severe malaria. Axillary temperature >= 37.5 ºC. Absence of signs of severe malnutrition. Absence of any obvious cause of fever other than malaria. No history of allergy to CQ. Willingness to return to the health facility for follow-up. Informed consent obtained from the caretaker of the child

Exclusion Criteria:

Danger signs of severe or complicated malaria, persisted vomiting. Received treatment with an antimalarial drug other than CQ in the last 2 weeks. Caretaker did not sign the consent form

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1035
Dates: Start 2002-07; Study Completion 2002-12

PRIMARY OUTCOMES:
Clinical and parasitological failure rates by day 14
Prevalence of pfcrt-76T, pfmdr1-86Y before treatment

SECONDARY OUTCOMES:
Proportion of children who cleared parasites carrying pfcrt-76T and pfmdr1-86Y alleles.
Prevalence of dhfr-51, 59, 108 and dhps-437, 540

CONTACTS AND LOCATIONS:
Overall Officials: Simon Cousens, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Brian M Greenwood, FRCP FRS, Principal Investigator — London School of Hygiene and Tropical Medicine; Diadier Diallo, MsC, Principal Investigator — Centre national de recherche et de formation sur le paludisme; Colin Sutherland, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Kadiogo, Burkina Faso